CLINICAL TRIAL: NCT02669628
Title: Anti-mullerian Hormone in Ovarian Reserve Evaluation After Treatment of Endometriomas With Alcohol Sclerotherapy Versus Surgery. A Pilot Study.
Brief Title: Antimullerian Hormone in Endometriomas
Status: Completed | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Roche Diagnostic Ltd. (Industry)
Responsible Party: Principal Investigator, Amparo Garcia-Tejedor, Dr, Hospital Universitari de Bellvitge
Other Study IDs: PR314/15
Record Dates: First submitted 2016-01-23; First posted 2016-02-01 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Endometriomas
MeSH Terms: conditions — Endometriosis | interventions — Wound Closure Techniques; Ethanol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical technique: Laparoscopic ovarian cystectomy
  Interventions: Procedure: Surgical technique
- Alcohol sclerotherapy: US-aspiration and alcohol sclerosis
  Interventions: Procedure: Alcohol sclerotherapy

INTERVENTIONS:
Procedure: Surgical technique — Laparoscopic surgery
  Groups: Surgical technique
Procedure: Alcohol sclerotherapy — US-guided sclerotherapy
  Groups: Alcohol sclerotherapy

SUMMARY:
The purpose of this multicenter study is to evaluate the ovarian reserve after alcohol sclerotherapy of endometriomas versus conventional surgery.

DETAILED DESCRIPTION:
Between 5-10% fertile women are affected by endometriosis, and ovarian endometrioma is present in 17-44% of cases, with 40% of patients with endometriomas being sterile. However, the "gold standard" treatment is laparoscopic ovarian cystectomy and this therapy is associated with a diminished ovarian reserve, with a significant antimullerian hormone (AMH) decrease.

Alcohol sclerotherapy is a new minimal invasive procedure in endometrioma treatment whose potential beneficial effect in fertility preservation is not still demonstrated.

The investigators would like to demonstrate that this procedure improves fertility preservation and reduces morbidity and costs in contrast with conventional surgery. Moreover,the investigators would like to demonstrate that this procedure could be performed in different centers with similar results.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age ≥18 and <40 years
* Unilocular endometrioma according ultrasounds
* Endometrioma size: 35-100 mm during > 3 months from diagnosis
* CA125 <200 IU/mL and HE4 < 70,
* AMH previous surgery between 1.2-4 ng/mL

Exclusion Criteria:

* Previous ovarian surgery or gynecological cancer
* Severe extraovarian endometriosis
* Dermoid or high risk of malignancy cysts
* Hormonal treatment 3 months before
* Pregnancy
* Mental disability

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with ultrasound suspicion of ovarian endometrioma (4-10 cm)
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
AMH Test | 6 months
  the value of AMH after both procedures in ng/mL

SECONDARY OUTCOMES:
antral follicles count | 6 months
  US antral follicles count after both procedures
tumoral markers: epididimal human protein 4 (HE-4) and CA125 | 6 months
  the value tumoral markers after both procedures
complications | 1 day
  number of participants with complications
costs | 1 day
  costs (euros) of the procedures and their complications

CONTACTS AND LOCATIONS:
Overall Officials: Amparo Garcia-Tejedor, MDPhD, Principal Investigator — Hospital de Bellvitge. IDIBELL
Locations (1):
- Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data should be available 6 months after the procedure

REFERENCES:
- [Background] Coccia ME, Rizzello F, Cammilli F, Bracco GL, Scarselli G. Endometriosis and infertility Surgery and ART: An integrated approach for successful management. Eur J Obstet Gynecol Reprod Biol. 2008 May;138(1):54-9. doi: 10.1016/j.ejogrb.2007.11.010. Epub 2008 Feb 20. PMID 18243485
- [Background] Muzii L, Bianchi A, Croce C, Manci N, Panici PB. Laparoscopic excision of ovarian cysts: is the stripping technique a tissue-sparing procedure? Fertil Steril. 2002 Mar;77(3):609-14. doi: 10.1016/s0015-0282(01)03203-4. PMID 11872220
- [Background] Raffi F, Metwally M, Amer S. The impact of excision of ovarian endometrioma on ovarian reserve: a systematic review and meta-analysis. J Clin Endocrinol Metab. 2012 Sep;97(9):3146-54. doi: 10.1210/jc.2012-1558. Epub 2012 Jun 20. PMID 22723324
- [Background] Biacchiardi CP, Piane LD, Camanni M, Deltetto F, Delpiano EM, Marchino GL, Gennarelli G, Revelli A. Laparoscopic stripping of endometriomas negatively affects ovarian follicular reserve even if performed by experienced surgeons. Reprod Biomed Online. 2011 Dec;23(6):740-6. doi: 10.1016/j.rbmo.2011.07.014. Epub 2011 Jul 27. PMID 22019621
- [Background] Akamatsu N, Hirai T, Masaoka H, Sekiba K, Fujita T. [Ultrasonically guided puncture of endometrial cysts--aspiration of contents and infusion of ethanol]. Nihon Sanka Fujinka Gakkai Zasshi. 1988 Feb;40(2):187-91. Japanese. PMID 3283269
- [Background] Noma J, Yoshida N. Efficacy of ethanol sclerotherapy for ovarian endometriomas. Int J Gynaecol Obstet. 2001 Jan;72(1):35-9. doi: 10.1016/s0020-7292(00)00307-6. PMID 11146075
- [Background] Messalli EM, Cobellis G, Pecori E, Pierno G, Scaffa C, Stradella L, Cobellis L. Alcohol sclerosis of endometriomas after ultrasound-guided aspiration. Minerva Ginecol. 2003 Aug;55(4):359-62. PMID 14581861
- [Background] Kafali H, Eser A, Duvan CI, Keskin E, Onaran YA. Recurrence of ovarian cyst after sclerotherapy. Minerva Ginecol. 2011 Feb;63(1):19-24. PMID 21311417
- [Background] Yazbeck C, Madelenat P, Ayel JP, Jacquesson L, Bontoux LM, Solal P, Hazout A. Ethanol sclerotherapy: a treatment option for ovarian endometriomas before ovarian stimulation. Reprod Biomed Online. 2009 Jul;19(1):121-5. doi: 10.1016/s1472-6483(10)60055-7. PMID 19573300
- [Background] Garcia-Tejedor A, Castellarnau M, Ponce J, Fernandez ME, Burdio F. Ethanol sclerotherapy of ovarian endometrioma: a safe and effective minimal invasive procedure. Preliminary results. Eur J Obstet Gynecol Reprod Biol. 2015 Apr;187:25-9. doi: 10.1016/j.ejogrb.2015.02.004. Epub 2015 Feb 16. PMID 25739052
- [Background] Somigliana E, Berlanda N, Benaglia L, Vigano P, Vercellini P, Fedele L. Surgical excision of endometriomas and ovarian reserve: a systematic review on serum antimullerian hormone level modifications. Fertil Steril. 2012 Dec;98(6):1531-8. doi: 10.1016/j.fertnstert.2012.08.009. Epub 2012 Sep 10. PMID 22975114
- [Background] Koike T, Minakami H, Motoyama M, Ogawa S, Fujiwara H, Sato I. Reproductive performance after ultrasound-guided transvaginal ethanol sclerotherapy for ovarian endometriotic cysts. Eur J Obstet Gynecol Reprod Biol. 2002 Oct 10;105(1):39. doi: 10.1016/s0301-2115(02)00144-6. PMID 12270563